CLINICAL TRIAL: NCT04687228
Title: Evaluating Body Acceptance Programs for Young Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Michael and Arlene Rosen Foundation (Unknown)
Responsible Party: Principal Investigator, Tiffany Brown, Principal Investigator & Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 201229S
Record Dates: First submitted 2020-12-15; First posted 2020-12-29 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Body Image Disturbance; Eating Disorder Symptom; Dysmorphia; Eating Disorders
Keywords: Male; Muscularity Oriented Eating; Exercise; Eating Disorder; Body Image
MeSH Terms: conditions — Congenital Abnormalities; Feeding and Eating Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will briefly be screened for eligibility criteria by phone. Eligible participants will be assessed using two structured clinical interviews (SCID-5 & EPSI-CRV) and complete a set of self-report measures at baseline. Following assessment participants will be randomized into one of two groups. One group will receive a dissonance-based intervention known as the More than Muscles (MTM), while other participants will engage in a Media Advocacy (MA) active control. Participants will complete the same set of self-report measures from baseline, after their final group, at 1-month follow-up and at 6-month follow-up. During the 6-month follow-up participants will also be reassessed using the same structured clinical interviews at baseline.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will remain unaware of what group they have been randomized to as both groups will be actively be participating in groups focused on male body image.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Media Advocacy (MA) (Active Comparator): Participants assigned to this condition take place in a time and attention-matched active control where they discuss the role of media in promoting the body ideal.
  Interventions: Behavioral: Media Advocacy (MA)
- Body Project: More than Muscles (MTM) (Experimental): Participants assigned to this condition take part in a two-session intervention based on dissonance theory which encourages them to challenge the body ideal.
  Interventions: Behavioral: More than Muscles (MTM)

INTERVENTIONS:
Behavioral: More than Muscles (MTM) — In session 1, the primary activities are: 1) define the "ideal" body type for men in our culture, 2) discuss the origin and perpetration of the "ideal," 3) brainstorm the costs of pursuing the "ideal," 4) participate in a verbal challenge during which participants counter the "ideal" message, and (5) are asked to complete three "homework" assignments (i.e., a letter to an adolescent boy, a behavioral challenge, and a mirror exposure assignment). In session 2, the primary activities are: 1) reviewing homework, 2) engage in role-plays to counter/discourage pursuit of the "ideal," 3) discuss ways to challenge and avoid "negative body talk" statements, 4) list ways to resist the pressure to pursue this "ideal" both individually and as a group within the larger community (i.e., body activism), 5) discuss barriers to body activism and strategies to overcome those barriers, and 6) individually select an exit exercise to continue to actively challenge the appearance ideal.
  Other Names: Body Project
  Arms: Body Project: More than Muscles (MTM)
Behavioral: Media Advocacy (MA) — MA content generally centers on acknowledging and discussing the role the media has on shaping body image ideals. Session 1: In session 1, similar to MTM, the primary activities will include: (1) describing the ideal body for men in our culture, (2) discussing how the media impacts this ideal, with a particular focus on advertising. Following this, participants will (3) watch a video on how the media influences body image among men, and the consequences of internalizing these messages. Session 2: In session 2, content will continue by further discussion of the video showed in session 1, with participants sharing their reactions. Next, the group discusses the attainability of the ideal as well as discusses other forms of media (e.g., social media) and how it impacts body image.
  Arms: Media Advocacy (MA)

SUMMARY:
While eating disorders in males are often overlooked, up to 7 million men in the United States will experience an Eating Disorder in their lifetime. Critically, men are less likely to seek treatment for an Eating Disorder compared to females. Therefore, prevention programs that target male-specific Eating Disorder risk factors prior to the development of an eating or appearance-related disorder are crucial in reducing eating disorders in this population. Preliminary work by our group established the initial efficacy of a novel program, the Body Project: More than Muscles (MTM) compared to assessment-only control. This study will replicate and extend this research by comparing MTM to a time and attention-matched control used in previous eating disorder prevention work, media advocacy (MA).

DETAILED DESCRIPTION:
Although often overlooked, Eating Disorders in men are a serious and deadly public health problem, affecting up to 7 million men in the United States. Efficacious, promulgated Eating Disorder treatments largely remain unknown, particularly for males. Over recent decades, men have faced increasing social pressures to obtain an unrealistically lean and muscular physique, which have contributed to body dissatisfaction and unhealthy eating and weight control behaviors among men, including symptoms of both Eating Disorders and muscle dysmorphia (body image disturbance characterized by the unhealthy pursuit of muscularity. Despite the impairment and distress associated with these conditions, males are less likely to seek treatment than females, in part due to stigma. Importantly, for those men who do seek help, existing treatments are targeted mostly towards females, rarely address male-specific risk factors, and are ineffective for over 50% of patients. Thus, well-accepted, easily replicable preventative programs that target male-specific Eating Disorder risk factors prior to disorder onset are critical to reduce the public health burden and disparities associated with eating disorders in men.

Research supports that for men, pressures from media, friends, partners, and family to pursue a lean, muscular body can lead to body-ideal internalization -- the belief that one's self-worth and value are defined by physical appearance. This can lead to dissatisfaction with muscularity and body fat, which in turn, contributes to eating disorder and muscle dysmorphia-related attitudes and behaviors. Thus, targeting internalization of the lean, muscular ideal portrayed in media culture would be important for reducing both Eating Disorder and muscle dysmorphia symptoms for men.

While studies have targeted body-ideal internalization in groups of women using dissonance-based interventions, until recently, no programs had been developed to address internalization of the lean, muscular body ideal for men. Our group recently developed and evaluated the Body Project: More than Muscles (MTM) in a randomized controlled trial (RCT) to target eating disorder and muscle dysmorphia risk factors in body-dissatisfied men. Results demonstrated significantly greater decreases in body-ideal internalization, dietary restraint, drive for muscularity, bulimic symptoms (e.g., binge eating, self-induced vomiting, laxatives, fasting, and/or excessive exercise), and muscle dysmorphia symptoms for men in the MTM intervention compared to assessment-only controls, both pre- to post-intervention and at 1-month follow-up. Further, body-ideal internalization mediated intervention outcomes for bulimic and muscle dysmorphia symptoms, supporting that the intervention's effects were exerted through reducing internalization of lean, muscular ideal images portrayed in media.

While initial results for MTM are promising, prior to disseminating this program to a wider audience, the present study will replicate and extend effects observed in the previous trial by comparing the intervention to a time- and attention-matched media advocacy (MA) active control condition used in previous Eating Disorder prevention programs. The present study will also explore the impact of MTM on additional risk factors for Eating Disorders and muscle dysmorphia in men not explicitly included in the previous RCT including unhealthy exercise, self- and other-objectification, appearance- and performance-enhancing drug (APED) use, and overall levels of depression, stress, and anxiety.

Results from the present study will provide critical support to help translate research on Eating Disorders and muscle dysmorphia in men into evidence-based prevention of these problems. MTM represents a novel approach to eating disorder prevention in this underserved population. This intervention has potential for wide dissemination, as peer-led interventions in women have demonstrated comparable impact to professional-led interventions. Further, if effects for MTM replicate, future research could adapt online or web-based versions of the program to help disseminate this program to a wider audience of men across the country. Thus, if results support the intervention's efficacy, this could lead to the expanded delivery of the intervention into university-based or online effectiveness trials to help prevent Eating Disorders and reduce body dissatisfaction for men at a national level.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 30 years old
* Identify as male
* Endorse body image concerns
* Speak English and able to provide informed consent

Exclusion Criteria:

* Diagnosis of a DSM-5 eating disorder determined by SCID-5
* Significant neuropsychiatric illness (e.g., dementia, untreated severe psychiatric illness determined by SCID-unmedicated bipolar disorder, psychosis, or active suicidal ideation)
* Older than 30 years old
* Younger than 18 years old

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Person who self-identify as male.
Enrollment: 137 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Examination Questionnaire (EDE-Q) | change from baseline to immediately post-intervention, change from baseline to 1-month follow-up, and change from baseline to 6-month follow-up
  The EDE-Q is a 28-item measure scored on a 7-point rating scale with scores ranging from 0 to 168 (scores higher than 4 on individual questions are indicative of clinical levels). The EDE-Q is a transdiagnostic measure of Eating Disorder symptoms with high scores indicating elevated eating pathology.
Muscle Dysmorphic Disorder Inventory (MDDI) | change from baseline to immediately post-intervention, change from baseline to 1-month follow-up, and change from baseline to 6-month follow-up
  The MDDI is a 13-item measure for muscle dysmorphia symptoms, which is a common feature of Eating Disorders in men. Items are scored 0 (never) to 4 (always) with higher scores indicating greater muscle dysmorphic symptoms. Scores on this measure range 0 to 52.
Eating Pathology Symptom Inventory-Clinician Rated Version (EPSI-CRV) | Change from baseline to 6-month follow-up related to dimensional changes in Eating Disorder-related psychopathology.
  The EPSI-CRV is a semi-structured interview that assesses dimensional constructs of psychopathology associated with Diagnostic and Statistical Manual-5 Eating Disorders. The interview will take approximately 40 minutes to complete.

SECONDARY OUTCOMES:
Sociocultural Attitudes Towards Appearance Questionnaire (SATAQ) | change from baseline to immediately post-intervention, change from baseline to 1-month follow-up, and change from baseline to 6-month follow-up
  The SATAQ is a 30-item measure of westernized beauty standards represented in media. Items are rated 1 (definitely disagree) to 5 (definitely agree) with scores ranging from 30 to 150. Higher scores indicate greater endorsement of beauty ideals portrayed in the media.
Drive for Muscularity Scale (DMS) | change from baseline to immediately post-intervention, change from baseline to 1-month follow-up, and change from baseline to 6-month follow-up
  The DMS is a 15-item measure of self-perceived muscularity. The measure utilizes a 6 point scale, (1) indicating always, and (6) denoting never. Lower scores indicate higher drive for muscularity. Scores range from 16 to 90 on the DMS.
Male Body Attitudes Scale (MBAS) | change from baseline to immediately post-intervention, change from baseline to 1-month follow-up, and change from baseline to 6-month follow-up
  The MBAS is a 29-item dimensional assessment of men's body attitudes. Items are scored from 1 (never) to 6 (always) with higher scores reflecting elevated negative body attitudes. Scores from this measure range from 29 to 174.
Self-Objectification Questionnaire (SOQ) | change from baseline to immediately post-intervention, change from baseline to 1-month follow-up, and change from baseline to 6-month follow-up
  The SOQ is a 20-item measure of how individuals appraise attributes in reference to themselves and their partner. Half of the questions relate to personal attributes the other half relate to a potential partners. The measure requires participants to rank the ten questions related to their personal attributes from 0 (least impact) to 9 (highest impact) and repeat the procedure for a potential partner.
Obligatory Exercise Questionnaire (OEQ) | change from baseline to immediately post-intervention, change from baseline to 1-month follow-up, and change from baseline to 6-month follow-up
  The OEQ is a 20-item measure of maladaptive exercise, a common feature in Eating Disorders. Responses are captured using a 4-point scale, 1 (never) to 4 (always), with higher scores indicating increased dysregulation relating to exercise. Scores range from 20 to 80 for this measure.
Appearance and Performance Enhancing Drug Use (APED; questions were derived from the Adolescents Training and Learning to Avoid Steroids [ATLAS] study) | change from baseline to immediately post-intervention, change from baseline to 1-month follow-up, and change from baseline to 6-month follow-up
  APED use was measured using 8-items derived from the ATLAS study. Participants are asked to respond from 1 (strongly agree) to 7 (strongly disagree) on the first 5 questions. Higher scores indicate elevated risk for future steroid use. The final 3-items request participants indicate if they have used anabolic steroids in the past 3 months (yes or no); if they have used supplements to alter their physical appearance (yes or no); if they answered yes to using supplements to alter their physical appearance, they were asked to endorse what specific substance was used (e.g., protein powder, creatine, testosterone booster, and fat burners).
Depression, Anxiety, Stress Scale (DASS-21) | change from baseline to immediately post-intervention, change from baseline to 1-month follow-up, and change from baseline to 6-month follow-up
  The DASS-21 is a 21-item measure that examines symptoms related to stress, anxiety, and depression. Participants are asked for respond on a scale from 0 (doesn't apply to me at all) to 3 (applies to me very much, or most of the time). Higher scores on the three sub-scales indicate elevated symptoms associated with depression, anxiety, or stress. Total scores range from 0 to 63. Each sub-scale is scored from 0 to 21.
Difficulties in Emotion Regulation Scale (DERS) short form | change from baseline to immediately post-intervention, change from baseline to 1-month follow-up, and change from baseline to 6-month follow-up
  The DERS-16 is a validated brief version of the original DERS (36-item measure). The brief version of the DERS, is a 16-item measure for dimensions of emotion dysregulation. Participants indicate how often each statement applies to them on a scale from 1 (almost never) to 5 (almost always). Scores for the measure range from 16 to 80, with higher scores indicating greater emotion regulation difficulty.
Acceptance and Action Questionnaire 2 (AAQ-II) | change from baseline to immediately post-intervention, change from baseline to 1-month follow-up, and change from baseline to 6-month follow-up
  The AAQ-II is a 7-item measure of experiential avoidance and psychological flexibility. Participants use a 7-point scale ranging from 1 (never true) to 7 (always true) in response to each statement. Scores range from 7 to 49, with higher scores indicating greater psychological inflexibility and avoidance of emotional experiences.
Intervention Acceptability | Immediately post-intervention
  Participants will respond to a 13-item measure of intervention acceptability for the MTM condition and MA condition. The first 10-items are scored on a 5 point scale, 1 indicating strongly disagree and 5 indicating strongly agree (higher score indicating higher acceptability). The last 3-items request participants provide written feedback about the intervention they participated in: which part of the program was most helpful? Which activity was the least helpful? Do you have any suggestions for improving the program? The last 3-items are not scored or included in the overall treatment acceptability score.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, Eating Disorder Center for Treatment and Research, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Principal Investigator will comply with data storage and sharing guidelines associated with her institutions best practices. Participant information will be de-identified in cases of sharing to maintain anonymity.

REFERENCES:
- [Background] Strother E, Lemberg R, Stanford SC, Turberville D. Eating disorders in men: underdiagnosed, undertreated, and misunderstood. Eat Disord. 2012;20(5):346-55. doi: 10.1080/10640266.2012.715512. PMID 22985232
- [Background] Hudson JI, Hiripi E, Pope HG Jr, Kessler RC. The prevalence and correlates of eating disorders in the National Comorbidity Survey Replication. Biol Psychiatry. 2007 Feb 1;61(3):348-58. doi: 10.1016/j.biopsych.2006.03.040. Epub 2006 Jul 3. PMID 16815322
- [Background] Keel PK. Eating Disorders. Upper Saddle River: Prentice Hall; 2005
- [Background] Kirkbride J, Coid JW, Morgan C, Fearon P, Dazzan P, Yang M, Lloyd T, Harrison GL, Murray RM, Jones PB. Translating the epidemiology of psychosis into public mental health: evidence, challenges and future prospects. J Public Ment Health. 2010 Jun;9(2):4-14. doi: 10.5042/jpmh.2010.0324. PMID 21160544
- [Background] Rodgers RF, Ganchou C, Franko DL, Chabrol H. Drive for muscularity and disordered eating among French adolescent boys: a sociocultural model. Body Image. 2012 Jun;9(3):318-23. doi: 10.1016/j.bodyim.2012.03.002. Epub 2012 Apr 10. PMID 22494958
- [Background] Tylka TL. Refinement of the tripartite influence model for men: dual body image pathways to body change behaviors. Body Image. 2011 Jun;8(3):199-207. doi: 10.1016/j.bodyim.2011.04.008. Epub 2011 Jun 12. PMID 21664886
- [Background] Litt D, Dodge T. A longitudinal investigation of the Drive for Muscularity Scale: predicting use of performance enhancing substances and weightlifting among males. Body Image. 2008 Dec;5(4):346-51. doi: 10.1016/j.bodyim.2008.04.002. Epub 2008 Jul 21. PMID 18644753
- [Background] Leit RA, Gray JJ, Pope HG Jr. The media's representation of the ideal male body: a cause for muscle dysmorphia? Int J Eat Disord. 2002 Apr;31(3):334-8. doi: 10.1002/eat.10019. PMID 11920996
- [Background] Cafri G, Thompson JK, Ricciardelli L, McCabe M, Smolak L, Yesalis C. Pursuit of the muscular ideal: Physical and psychological consequences and putative risk factors. Clin Psychol Rev. 2005 Feb;25(2):215-39. doi: 10.1016/j.cpr.2004.09.003. Epub 2004 Dec 30. PMID 15642647
- [Background] Pope HG Jr, Gruber AJ, Choi P, Olivardia R, Phillips KA. Muscle dysmorphia. An underrecognized form of body dysmorphic disorder. Psychosomatics. 1997 Nov-Dec;38(6):548-57. doi: 10.1016/S0033-3182(97)71400-2. PMID 9427852
- [Background] Olivardia R, Pope HG Jr, Hudson JI. Muscle dysmorphia in male weightlifters: a case-control study. Am J Psychiatry. 2000 Aug;157(8):1291-6. doi: 10.1176/appi.ajp.157.8.1291. PMID 10910793
- [Background] Bramon-Bosch E, Troop NA, Treasure JL. Eating disorders in males: a comparison with female patients. European Eating Disorders Review. 2000;8(4):321-328.
- [Background] Griffiths S, Hay P, Mitchison D, Mond JM, McLean SA, Rodgers B, Massey R, Paxton SJ. Sex differences in the relationships between body dissatisfaction, quality of life and psychological distress. Aust N Z J Public Health. 2016 Dec;40(6):518-522. doi: 10.1111/1753-6405.12538. Epub 2016 Jul 3. PMID 27372301
- [Background] Griffiths S, Mond JM, Li Z, Gunatilake S, Murray SB, Sheffield J, Touyz S. Self-stigma of seeking treatment and being male predict an increased likelihood of having an undiagnosed eating disorder. Int J Eat Disord. 2015 Sep;48(6):775-8. doi: 10.1002/eat.22413. Epub 2015 Jun 6. PMID 26052695
- [Background] Striegel-Moore RH, Leslie D, Petrill SA, Garvin V, Rosenheck RA. One-year use and cost of inpatient and outpatient services among female and male patients with an eating disorder: evidence from a national database of health insurance claims. Int J Eat Disord. 2000 May;27(4):381-9. doi: 10.1002/(sici)1098-108x(200005)27:43.0.co;2-u. PMID 10744844
- [Background] Brown TA, Keel PK. Current and emerging directions in the treatment of eating disorders. Subst Abuse. 2012;6:33-61. doi: 10.4137/SART.S7864. Epub 2012 Mar 29. PMID 22879753
- [Background] Keel PK, Brown TA. Update on course and outcome in eating disorders. Int J Eat Disord. 2010 Apr;43(3):195-204. doi: 10.1002/eat.20810. PMID 20186717
- [Background] Pope HG Jr, Olivardia R, Gruber A, Borowiecki J. Evolving ideals of male body image as seen through action toys. Int J Eat Disord. 1999 Jul;26(1):65-72. doi: 10.1002/(sici)1098-108x(199907)26:13.0.co;2-d. PMID 10349585
- [Background] Leit RA, Pope HG Jr, Gray JJ. Cultural expectations of muscularity in men: the evolution of playgirl centerfolds. Int J Eat Disord. 2001 Jan;29(1):90-3. doi: 10.1002/1098-108x(200101)29:13.0.co;2-f. PMID 11135340
- [Background] Pope H, Phillips KA, Olivardia R. The Adonis complex: The secret crisis of male body obsession: Simon and Schuster; 2000.
- [Background] Harrison K, Cantor J. The relationship between media consumption and eating disorders. Journal of communication. 1997;47(1):40-67.
- [Background] Brown TA, Forney KJ, Pinner D, Keel PK. A randomized controlled trial of The Body Project: More Than Muscles for men with body dissatisfaction. Int J Eat Disord. 2017 Aug;50(8):873-883. doi: 10.1002/eat.22724. Epub 2017 May 8. PMID 28481431
- [Background] Becker CB, Smith LM, Ciao AC. Peer-facilitated eating disorder prevention: A randomized effectiveness trial of cognitive dissonance and media advocacy. Journal of Counseling Psychology. 2006;53(4):550.
- [Background] Becker CB, Bull S, Schaumberg K, Cauble A, Franco A. Effectiveness of peer-led eating disorders prevention: a replication trial. J Consult Clin Psychol. 2008 Apr;76(2):347-54. doi: 10.1037/0022-006X.76.2.347. PMID 18377130
- See also: Lab Website — https://brownlabucsd.wixsite.com/ucsdbodyacceptance